CLINICAL TRIAL: NCT05073055
Title: Comparison of Spinal Anesthesia and Erector Spina Plane Block in Unilateral Inguinal Hernias: A Randomized Controlled Study
Brief Title: Spinal Anesthesia Versus Erector Spina Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Mustafa Kaçmaz, Anesthesiology department director, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/38
Record Dates: First submitted 2021-03-22; First posted 2021-10-11 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Inguinal Hernia Repair; Postoperative Pain; Peripheral Nerve Blocks
Keywords: nerve block; inguinal hernia; anesthesia; spinal
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Spinal anesthesia was determined as the standard method. Erectile spina block was determined as a research group. There were equal numbers of patients in both groups. The patients to be assigned to the groups were determined by the closed envelope drawing method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SA (Active Comparator): Group 1 (SE) (n = 35): patients undergoing spinal anesthesia of patients in our hospital to do unilateral inguinal hernia operation. Block application and the times when the sensory block reaches the T10 level are recorded. Surgery is allowed in patients who develop sensory block at the T10 level. During our study, no changes will be made to the procedure described above, which is standardized during our study, only patient data will be recorded observationally. Patients who do not have sufficient sensory block to start the procedure despite waiting 10 minutes will be registered and excluded from the study and additional anesthesia will be applied.
  Interventions: Procedure: İnguinal Hernia Repair
- Group ESP+TA (Active Comparator): Group 2 (Errector spina block + TA) (n = 35): 2% lidocaine hydrochloride (10 mg / ml) 15 ml, 0.5% bupivacaine hydrochloride (20 mg / ml) 15 ml, serum 8.4% Sodium Bicarbonate 5 ml to be used for each patient before the operation in order to apply the erectile spina block block with tumescent anesthesia. Adding adrenaline tartrate (5 μg / mL) to 5 ml with saline, a total of 40 ml of mixture was prepared. Hydrodissection was achieved using a 5 cm, 21G peripheral nerve block needle just below the erector spina muscle on the Transverse Process of L1. Afterwards, a unilateral injection of 15 ml at T12 and L1 levels was applied to each segment with the needle directed at two different angles from the same insertion point.
  Interventions: Procedure: İnguinal Hernia Repair

INTERVENTIONS:
Procedure: İnguinal Hernia Repair — After hemodynamic stability, the patient was placed in the lateral position and infiltration anesthesia with 2% lidocaine was applied. Following aseptic preparation of the skin and probe, a medium-frequency curvey USG transducer was first placed in the midline to visualize the transverse projection of the first lumbar (L1) vertebra, then moved 2.5 cm laterally in the parasagittal plane, after imaging the transverse process, in-plane spreading was injected. Hydrodissection was achieved on the TP of L1 by using a 5 cm, 21G peripheral nerve block needle just below the erector spina muscle with real-time imaging of the substance. Afterwards, a unilateral injection of 15 ml at T12 and L1 levels was applied to each segment with the needle directed at two different angles from the same insertion point.
  Other Names: Erectör spinae block; Spinal Anesthesia

SUMMARY:
The primary aim of our study was to use spinal anesthesia for unilateral inguinal hernia surgery and lumbar erector spina block supported by local infiltration anesthesia in terms of operation time, intraoperative hemodynamic data, motor block onset time, block termination time, analgesic need, discharge time, patient satisfaction, surgeon satisfaction. is to compare. Its second purpose is to observe nausea, vomiting, urinary retention, headache, chills, bleeding, wound infection.

DETAILED DESCRIPTION:
Seventy cases of the American Society of Anesthesia physical status (ASA) I-III class between the ages of 18-75 who were hospitalized in the general surgery clinic with the diagnosis of unilateral inguinal hernia will be enrolled in this study prospectively and randomly. The entire work will be conducted in accordance with the principles of the Declaration of Helsinki. The patients will be determined one day in advance with the single-blind method and the closed envelope method, and all patients will be informed about the study plan in detail, and informed patient consent will be obtained.

Patients with liver disease, allergy to anesthetic agents, local infection, recurrence, strangulated hernia, patients with a history of allergy to local anesthetics, and patients with a history of anesthesia up to two weeks ago will be excluded from the study. The general surgeon who performs the inguinal hernia repair surgery will not take part in the postoperative follow-up of the patients. Patients with a diagnosis of inguinal hernia who are operated on in our hospital are administered 0.1 mg.kg-midazolam 30 minutes before the block application. Electrocardiogram (ECG), heart rate (HR), peripheral oxygen saturation (SpO2) are monitored in the pre-anesthesia preparation room, and nasal hydration application with 2 l / min O2 and 5 ml kg hr, 0.9% NaCl is started. These patients will be randomly divided into two groups. Patients who underwent spinal anesthesia will be named as Group 1, and patients who underwent Erectile Spina Block and Tumescent anesthesia as Group 2.

Group 1 (SE) (n = 35): patients undergoing spinal anesthesia of patients in our hospital to do unilateral inguinal hernia operation, is taken to a seated position on the operating table and a 25 gauge spinal needle under sterile conditions (dominant, Turkey) subarachnoid space entered% in 30 seconds 0, 5 units of levobupivacaine 3 mL is injected. The intervention is started after the patients are placed in the supine position immediately after the spinal block and the level of the sensory block is confirmed by the pin prick test to be at the T10 dermatome. Block application and the times when the sensory block reaches the T10 level are recorded. Surgery is allowed in patients who develop sensory block at the T10 level. During our study, no changes will be made to the procedure described above, which is standardized during our study, only patient data will be recorded observationally. Patients who do not have sufficient sensory block to start the procedure despite waiting 10 minutes will be registered and excluded from the study and additional anesthesia will be applied.

Group 2 (Errector spina block + TA) (n = 35): To be used for each patient before the operation to apply tumescent anesthesia-assisted erectile spina block to patients undergoing unilateral inguinal hernia operation in our hospital with erectile spina block + infiltration anesthesia method. A total of 30 ml of mixture is prepared including lidocaine hydrochloride 10mg / ml, adrenaline tartarate (1: 1000) 5 μg / mL, 13 ml in total, 0.5% bupivacaine hydrochloride 13 ml, Sterile Serum 8.4% Sodium Bicarbonate 4 ml. After hemodynamic stability, the patient is placed in the lateral position and infiltration anesthesia with 2% lidocaine is applied. Following aseptic preparation of the skin and probe, a high-frequency linear USG transducer is moved 2.5 cm laterally in the parasagittal plane to visualize the transverse projection of the first lumbar (L1) vertebra. The needle, with real-time imaging of the spreading injected material, TP of L1 and at this level, just below the erector spina muscle, 5 cm, 21G peripheral nerve block needle (Pajuk®, stimuplex HNS12 Germany, Germany) is preferred. During the application, the needle is inserted perpendicular to the skin. Unilateral block is applied at T12 and L1 levels, with 10 ml in each segment. After the needle is withdrawn, pressure is applied to the injection area for 2 minutes and then, the patient is taken to the operation room, the prepared local anesthetic mixture is applied to the patient using the step-by-step technique, 5 ml under the skin and the subcutaneous area around the incision, and the other 5 ml under the fascia, the funiculus (spermatic cord). Tumescent anesthesia is applied around the area and the tissues at the base of the hernia sac. Surgery is permitted in patients who develop sensory block between T10-L1 dermatomes. In our study, patients whose sensory block is controlled by pin-prick test, and patients whose local anesthesia does not create sufficient sensory block to start the skin incision will be excluded from the study and additional anesthesia methods will be applied. The time during which the sensory blocks of the patients disappear will be recorded.

During surgery, the sedation level of the patients will be monitored with the Ramsey sedation score (1: agitated, anxiosis, 2: cooperative, 3: response to verbal commands, 4: vivid response to glabella hit or loud stimulus, 5: lazy response to glabella beat or loud stimulus, 6 : no answer).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inguinal hernia repair.
* Unilateral inguinal hernia.
* Patients with ASA II-III preoperative anesthesia score.

Exclusion Criteria:

* Patients with liver disease,
* allergy to anesthetic agents
* local infection,
* recurrence,
* strangulated hernia,
* patients with a history of allergy to local anesthetics,
* patients with a history of anesthesia up to two weeks ago

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Intraoperative pain score | 5 month
  The pain level felt by the patients during the operation will be measured using a visual analog scale. The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image.0 means being painless and 10 means the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa KAÇMAZ, Md, Study Director — Ömer Halisdemir Üniversity
Locations (1):
- Mustafa KAÇMAZ, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Group information, intraoperative and postoperative pain scores, amount of analgesic use, and length of stay in the hospital will be shared.

REFERENCES:
- [Result] Aksu C, Gurkan Y. Opioid sparing effect of Erector Spinae Plane block for pediatric bilateral inguinal hernia surgeries. J Clin Anesth. 2018 Nov;50:62-63. doi: 10.1016/j.jclinane.2018.06.048. Epub 2018 Jul 1. No abstract available. PMID 29980003
- [Result] Schwartzmann A, Peng P, Maciel MA, Forero M. Mechanism of the erector spinae plane block: insights from a magnetic resonance imaging study. Can J Anaesth. 2018 Oct;65(10):1165-1166. doi: 10.1007/s12630-018-1187-y. Epub 2018 Aug 3. No abstract available. PMID 30076575
- [Result] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771